CLINICAL TRIAL: NCT03215797
Title: Comparison of the Effects of Norepinephrine and Phenylephrine on Tissue Oxygenation and Hemodynamic Stability During an SVV Fluid Guided Therapy in Elderly Undergoing Radical Resection of Colon Cancer Surgery
Brief Title: Phenylephrine or Norepinephrine for a Better Hemodynamic Stability
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ph Vs N in SVV GDT
Record Dates: First submitted 2017-04-09; First posted 2017-07-12 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-04

CONDITIONS: Hypotension; Fluid Therapy
Keywords: svv; norepinephrine; phenylephrine; elderly
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Vasoconstrictor Agents; Norepinephrine; Catecholamines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phenylephrine and norepinephrine (Active Comparator): Phenylephrine 100ug/ml and Norepinephrine 5ug/ml IV infusion at a rate of 5 ml/h in case of perioperative hypotension.
  Interventions: Drug: phenylephrine; Drug: Norepinephrine
- Norepinephrine and phenylephrine (Other): Phenylephrine 100ug/ml and Norepinephrine 5ug/ml IV infusion in postoperative time in case of hypotension
  Interventions: Drug: phenylephrine; Drug: Norepinephrine

INTERVENTIONS:
Drug: phenylephrine — phenylephrine 100ug/ml IV infusion at a rate of 5ml/h in case of hypotension.
  Other Names: α1-adrenergic receptor agonist; vasopressor
Drug: Norepinephrine — Norepinephrine 5ug/ml IV infusion at a rate of 5 ml/h in case of hypotension
  Other Names: noradrenaline; catecholamine

SUMMARY:
A prospective, double-blinded study. The present study consisted in applying Stroke volume variation fluid guided therapy to old patients (65 years old) undergoing radical resection of colon surgery. The aim of this study is to compare the effects of norepinephrine and phenylephrine in treating perioperative hypotension, and to find the safest and most effective vasopressor for elderly.

DETAILED DESCRIPTION:
Fluid management has a great influence on patient's morbidity, mortality and on the overall outcome.Goal directed therapy was proved by multiple studies to be a goal therapy in maintaining a stable hemodynamic state. Nevertheless, as the population worldwide is aging, elderly presenting for surgery are also increasing. This population is known for the multiple comorbidities and physiological changes which makes them prone to dehydration and hypotension. That's when we are going to use either Norepinephrine in one group or Phenylephrine in the other and compare the effects of both vasopressors.

Parameters we are going to use are: Hemodynamic (HR, MAP, CO, CI, SVV, SV); Tissue Oxygenation and perfusion (DO2, VO2, ERO2, CRT, Lactate, blood gas); Urine output.

ELIGIBILITY:
Inclusion Criteria:

* Operation time should be equal or greater than 2h,
* Patients older than 65 years old,
* ASA Ⅱ or Ⅲ.

Exclusion Criteria:

* Clear arrhythmia,
* Need to apply PEEP,
* Peripheral vascular disease and arterial catheter contraindications.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
the tissue oxygenation | from the beginning of surgery to the end of surgery
  it means the tissue oxygen delivery and consumption

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-01-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT03215797/Prot_000.pdf